CLINICAL TRIAL: NCT00001020
Title: A Phase I Study of the Safety and Immunogenicity of rgp120/HIV-1IIIB Vaccine in Healthy Adult Subjects (NOTE: Study Extended ONLY for Subjects Who Have Previously Received rgp120/HIV-1IIIB or rgp120/HIV-1MN on VEU 006 or VEU 006 Rollover Study)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 006X; VEU 006; V0199g; 11537 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Viral Vaccines; HIV-1; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: rgp120/HIV-1IIIB
Biological: rgp120/HIV-1MN

SUMMARY:
AMENDED 11/17/93: To determine whether the pattern of response to MN rgp120 vaccine is altered by pre-exposure to IIIB rgp120.

ORIGINAL DESIGN: To evaluate the safety (clinical and immunologic) of rgp120/HIV-1IIIB vaccine (gp120 vaccine) immunization in healthy HIV-1 seronegative adult subjects. To compare the immune response to 100 mcg gp120 vaccine versus 300 mcg gp120 vaccine. To determine whether gp120 vaccine immunization causes a significant immune response as defined by specific parameters (e.g., induction of neutralizing antibodies to the IIIB isolate of HIV-1, gp120 antigen-specific lymphocytic proliferation).

Recent evidence suggests that gp120 is the HIV-1 protein with the greatest potential as a vaccine against HIV-1 infection. The gp120 envelope protein may be produced by recombinant DNA technology, and studies have shown that the vaccine is capable of eliciting neutralizing antibody activity in both rodents and nonhuman primate species.

DETAILED DESCRIPTION:
Recent evidence suggests that gp120 is the HIV-1 protein with the greatest potential as a vaccine against HIV-1 infection. The gp120 envelope protein may be produced by recombinant DNA technology, and studies have shown that the vaccine is capable of eliciting neutralizing antibody activity in both rodents and nonhuman primate species.

AMENDED 11/17/93: Selected subjects from VEU 006 or VEU 006 Rollover study will receive two injections of MN rgp120 vaccine, administered 28 days apart beginning 10-16 months after their last injection. Eight additional clinic visits will be required. Subjects are followed for at least 6 months.

ORIGINAL DESIGN: Twenty-eight subjects will be randomized to receive 100 or 300 mcg rgp120/HIV-1IIIB vaccine (gp120 vaccine) or matching placebo. For each dose level, 10 subjects will receive vaccine and four subjects will receive matching placebo. Injections are given intramuscularly at 0, 4, and 32 weeks. Each subject receiving treatment at the lower dose level must be monitored for unacceptable toxicity for at least 2 weeks following the initial immunization before his or her second dose is administered and before treatment at the higher dose level begins. Subjects are followed for at least 12 months.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV seronegativity.
* Good general health.
* No high-risk behavior for HIV infection.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Postive PPD (unless a chest x-ray is negative and there is no suggestion of active or old pulmonary tuberculosis).
* Positive VDRL or HBsAG.
* No febrile illness within 1 week of study.

Concurrent Medication:

Excluded:

* Concomitant corticosteroids or other known immunosuppressive drugs.
* Other experimental agents.

Patients with the following prior conditions are excluded:

* History of clinically significant cardiac, pulmonary, hepatic, renal, neurologic, or autoimmune disease.

Prior Medication:

Excluded:

* Other immunization within 4 weeks prior to study entry.

Identifiable high-risk behavior for HIV infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clements M, Study Chair; Belshe R, Study Chair
Locations (3):
- United States (3):
  - St Louis Univ School of Medicine, St Louis, Missouri
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington

REFERENCES:
- [Background] Clements ML, Belshe R, Duliege AM, Schwartz D, Gorse G, Izu A, Ammann A. Safety and immunogenicity of IIIB rgp120/HIV-1 vaccine in seronegative volunteers. The NIAID-sponsored AIDS Vaccine Clinical Trials Network. Int Conf AIDS. 1992 Jul 19-24;8(1):Mo9 (abstract no MoB 0026)
- [Background] Berman PW, Eastman DJ, Wilkes DM, Nakamura GR, Gregory TJ, Schwartz D, Gorse G, Belshe R, Clements ML, Byrn RA. Comparison of the immune response to recombinant gp120 in humans and chimpanzees. AIDS. 1994 May;8(5):591-601. doi: 10.1097/00002030-199405000-00004. PMID 7520248
- [Background] VanCott TC, Bethke FR, Burke DS, Redfield RR, Birx DL. Lack of induction of antibodies specific for conserved, discontinuous epitopes of HIV-1 envelope glycoprotein by candidate AIDS vaccines. J Immunol. 1995 Oct 15;155(8):4100-10. PMID 7561123
- [Background] Francis DP, Gregory T, McElrath MJ, Belshe RB, Gorse GJ, Migasena S, Kitayaporn D, Pitisuttitham P, Matthews T, Schwartz DH, Berman PW. Advancing AIDSVAX to phase 3. Safety, immunogenicity, and plans for phase 3. AIDS Res Hum Retroviruses. 1998 Oct;14 Suppl 3:S325-31. PMID 9814961
- [Background] Schwartz DH, Cosentino LM, Shirai A, Conover J, Daniel S, Klinman DM. Lack of correlation between the number of circulating B cells and the concentration of serum antibodies reactive with the HIV-1 envelope glycoprotein. J Acquir Immune Defic Syndr (1988). 1994 May;7(5):447-53. PMID 8158537
- [Background] Gorse GJ, Patel GB, Mandava M, Berman PW, Belshe RB. MN and IIIB recombinant glycoprotein 120 vaccine-induced binding antibodies to native envelope glycoprotein of human immunodeficiency virus type 1 primary isolates. National Institute of Allergy and Infectious Disease Aids Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1999 Jul 1;15(10):921-30. doi: 10.1089/088922299310638. PMID 10408729
- [Background] Schwartz DH, Gorse G, Clements ML, Belshe R, Izu A, Duliege AM, Berman P, Twaddell T, Stablein D, Sposto R, et al. Induction of HIV-1-neutralising and syncytium-inhibiting antibodies in uninfected recipients of HIV-1IIIB rgp120 subunit vaccine. Lancet. 1993 Jul 10;342(8863):69-73. doi: 10.1016/0140-6736(93)91283-r. PMID 8100910
- [Background] Gorse GJ, Patel GB, Newman FK, Belshe RB, Berman PW, Gregory TJ, Matthews TJ. Antibody to native human immunodeficiency virus type 1 envelope glycoproteins induced by IIIB and MN recombinant gp120 vaccines. The NIAID AIDS Vaccine Evaluation Group. Clin Diagn Lab Immunol. 1996 Jul;3(4):378-86. doi: 10.1128/cdli.3.4.378-386.1996. PMID 8807200